CLINICAL TRIAL: NCT01066975
Title: Mechanical Load on the Shoulders While Carrying a Backpack- Towards a Knowledge-Based Backpack Design
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Nogah Shabshin, Sheba Medical Center
Other Study IDs: SHEBA-10-7645-NS-CTIL
Record Dates: First submitted 2010-02-03; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Healthy; Strain
Keywords: loaded backpack; unloaded backpack
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- young and fit: 5 healthy subjects, age lower than 30 yrs and high physical fitness

SUMMARY:
Soldiers and recreational backpackers are often required to carry heavy loads on their body during military operations or hiking. Despite the advances in backpack design, the loads carried by soldiers still impose an extreme physiological strain (soft tissue deformation) which frequently results in discomfort, pain,musculoskeletal injuries, and loss sensorimotor function.

In the current study, characterization of the pressures, evaluation of the deformations of the soft tissues, specifically the fat, muscles, Brachial plexus and subclavian vessels applied on the shoulder while sitting with a heavy backpack will performed. The data acquired in the current trials will be used for development of a finite element (FE) 3D shoulder model. The purpose is to better understand the mechanical loads that are being transferred to the underlying tissue below the shoulder straps during walking/marching with a backpack. During the 2nd phase of this project, data collected during this research will be used to develop gear that will alleviate the strain on the shoulders, prevent injury, and enhance performance.

Hypothesis

* High focal strain (hot-spots) on the shoulder tissue that are observed with the pressure mapping will be observed also in the MR scans.
* The strain at those hot-spots can be reduced by personal-geometry adjusted straps.

Volunteers

Five young (18-30 yrs), healthy, and fit males will participate in this study.

Trials design

1. MR Scans- The scan will be performed for analysis of personal shoulder anatomy, and will be used for developing a 3D FE model. The sagittal view will be used to develop the 3D model. The coronal and axial sectional views will be used to assess the deformations applied on the shoulder tissue. The scan will then be repeated while carrying a 25 kg standard commercial backpack while sitting in the same position, for the assessment of shoulder girdle tissues deformations. Time estimation for each scan is 40 min (80 min total). The subjects are not required to carry the backpack prior to those scans.
2. Static pressure measurement- each volunteer will be asked to sit for 30 seconds while carrying the 25 kg backpack. During this session, pressure will be measured using a pressure mapping pad (Sensor Products Inc., USA) placed between the shoulder strap and the underlying tissue.

The maximal total participation time of each volunteer will be 2 hours total (inside and outside the MR).

Data acquired in the current trials will be used for the development of a FE (finite element) 3D shoulder model. MR scans will be utilized for composing geometry and for the boundary conditions assessment (strain magnitude). Pressure measurements will be used as boundary conditions (stress magnitude).

MR scans and pressure measurements will be performed in the Sheba medical center facilities.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 yrs
* healthy
* fit
* males

Exclusion Criteria:

* contraindications for MRI

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Five young (18-30 yrs), healthy, and fit males will participate in this study. Prior to signing a consent form, the PI will explain to the subjects about the MRI that they are about to participate in if they will decide to sign including all the discomforts involved in this study. For subjects that don't have contraindications for MRI there are no reported risks.
  The subjects will be informed that each one of them is free to decide, and is free to stop his participation any time he wishes to.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hadid, BSc, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel